CLINICAL TRIAL: NCT04129086
Title: Ketamine for Acute Pain After Trauma: KAPT Trial
Brief Title: Ketamine for Acute Pain Management After Trauma
Acronym: KAPT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, John Andrew Harvin, Associate Professor of Surgery, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSC-MS-19-0726
Record Dates: First submitted 2019-10-10; First posted 2019-10-16 (Actual); Results first posted 2023-04-21 (Actual); Last update posted 2023-04-21 (Actual); Status verified 2023-03

CONDITIONS: Trauma Injury; Pain; Opioid Use
Keywords: Multimodal Pain Therapy; Ketamine; Trauma
MeSH Terms: conditions — Accidental Injuries; Pain; Wounds and Injuries | interventions — Ketamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ketamine plus Usual care (Experimental)
  Interventions: Drug: Ketamine plus usual care
- Usual care (Active Comparator)
  Interventions: Drug: Usual Care

INTERVENTIONS:
Drug: Ketamine plus usual care — Bolus of .35 mg/kg Infusion start @ 0.15 mg/kg/hr; titrate range is 0.1 - 0.25 mg/kg/hr for 24 to 48 hours after admission and each subsequent major surgery plus multi-modal pain therapy considered as standard of care. Standard of care medications include Acetaminophen 1000 mg po q6 hours, Naproxen 500 mg po q12 hours, Gabapentin 300 mg po q8 hours and Lidocaine patch q 12 hours.
  Arms: Ketamine plus Usual care
Drug: Usual Care — Standard of care medications include Acetaminophen 1000 mg po q6 hours, Naproxen 500 mg po q12 hours, Gabapentin 300 mg po q8 hours and Lidocaine patch q 12 hours.
  Arms: Usual care

SUMMARY:
The purpose of this study is to compare the effectiveness of Ketamine drip along with usual care and usual care alone on trauma patients and to longitudinally quantify the pain experience of patients during hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* Adult trauma patients
* Admission to Shock Trauma ICU (STICU) or Surgical Intermediate Unit (SIMU)
* Randomization within 6 hours of arrival

Exclusion Criteria:

* Patient not expected to survive
* Contraindications to ketamine Allergy, Poorly controlled hypertension, Cardiac arrhythmia disorders (including atrial fibrillation), congestive heart failure, unstable coronary artery disease or recent myocardial infarction( MI)(within 6 months), cirrhosis, seizure disorder, and for those patients with unknown medical history - median sternotomy scar, mechanism of injury is fall from standing, 65 years of age or older, any arrhythmia on EKD)
* pregnancy
* in police custody
* history of dementia or movement disorder (i.e. Parkinson's)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2020-07-01 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John P Harvin, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Klugh JM, Puzio TJ, Wandling MW, Guy-Frank CJ, Green C, Sergot PB, Prater SJ, Balogh J, Stephens CT, Wade CE, Kao LS, Harvin JA. Ketamine for acute pain after trauma: A pragmatic, randomized clinical trial. J Trauma Acute Care Surg. 2024 Oct 1;97(4):514-519. doi: 10.1097/TA.0000000000004325. Epub 2024 May 1. PMID 38689402
- [Derived] Puzio TJ, Klugh J, Wandling MW, Green C, Balogh J, Prater SJ, Stephens CT, Sergot PB, Wade CE, Kao LS, Harvin JA. Ketamine for acute pain after trauma: the KAPT randomized controlled trial. Trials. 2022 Jul 27;23(1):599. doi: 10.1186/s13063-022-06511-6. PMID 35897081

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 305 were enrolled, but 5 did not consent to continue participation in the study.
Period: Overall Study
Arm/Group | Ketamine Plus Usual Care | Usual Care
Started | 144 | 156
Completed | 144 | 156
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine Plus Usual Care | Usual Care | Total
Number analyzed (Participants) | 144 | 156 | 300
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 34 [25 to 46] | 36 [27 to 50] | 35 [25 to 48]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28 | 36 | 64
  Male | 116 | 120 | 236
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 38 | 56 | 94
  Black | 39 | 56 | 95
  Hispanic | 59 | 41 | 100
  Other | 7 | 3 | 10
  Unknown | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 144 | 156 | 300
Number of Participants with Prior Opioid Use [Count of Participants; unit: Participants]
  No | 80 | 84 | 164
  Yes | 37 | 48 | 85
  Unknown | 27 | 24 | 51
Number of Participants with a History of Smoking [Count of Participants; unit: Participants]
  No | 73 | 84 | 157
  Yes | 48 | 52 | 100
  Unknown | 23 | 20 | 43
Number of Participants with a Positive Alcohol Screen [Count of Participants; unit: Participants]
  No | 85 | 91 | 176
  Yes | 35 | 37 | 72
  Not performed | 24 | 28 | 52
Number of Participants with a Positive Drug Screen [Count of Participants; unit: Participants]
  No | 41 | 62 | 103
  Yes | 61 | 51 | 112
  Not performed | 42 | 43 | 85

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Opioid Use as Measured by the Morphine Milligram Equivalents (MME) Per Day
Time Frame: In-hospital days (up to 6 weeks post hospital admission)
Measure: Mean (95% Confidence Interval); unit: MME per day
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 144 | 156
MME per day | 32 [29 to 36] | 39 [35 to 44]

2. Secondary Outcome: Pain as Assessed by Score on the Numeric Rating Scale (NRS)
Description: The NRS ranges from 0 (no pain) to 10 (worst pain), with a higher score indicating a worse outcome. This scale is used in verbal participants.
Time Frame: Hospital discharge (up to 6 weeks post hospital admission)
Population: Data were not collected for this outcome measure
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Patients That Showed Signs of Delirium During In-hospital Stay
Description: Incidence of delirium during in-hospital stay
Time Frame: Hospital discharge (up to 6 weeks post hospital admission)
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 144 | 156
Participants | 16 | 9

4. Secondary Outcome: Number of Patients That Required Unplanned Intubation During In-hospital Stay
Description: incidence of need for unplanned intubation during in-hospital stay
Time Frame: Hospital discharge (up to 6 weeks post hospital admission)
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 144 | 156
Participants | 2 | 3

5. Secondary Outcome: Number of Patients Who Required Unplanned Admission to Intensive Care Unit During In-hospital Stay
Description: Incidence of need for unplanned admission to an ICU
Time Frame: Hospital discharge (up to 6 weeks post hospital admission)
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 144 | 156
Participants | 7 | 7

6. Secondary Outcome: Initiation of Ketamine Drip
Description: Time from admission to time Ketamine drip started
Time Frame: Hospital discharge (up to 6 weeks post hospital admission)
Population: Data were not collected for this outcome measure
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Duration of Ketamine Drip
Description: Length of time Ketamine drip was infused
Time Frame: Hospital discharge (up to 6 weeks post hospital admission)
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 144 | 156
hours | 60 [32 to 86] | 76 [31 to 94]

8. Secondary Outcome: Number of Patients Requesting to Discontinue Ketamine
Description: Number of patients requesting to stop Ketamine for any complaint
Time Frame: Hospital discharge (up to 6 weeks post hospital admission)
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 144 | 156
Participants | 9 | 0

9. Secondary Outcome: Use of Other Pain Control Adjuncts Including Regional Anesthesia and Lidocaine Patch
Description: Incidence of use of additional pain control adjuncts such as regional anesthesia and lidocaine patch during hospitalization
Time Frame: Hospital discharge (up to 6 weeks post hospital admission)
Population: Lidocaine drip was not used in clinic.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 144 | 156
Participants
  Regional anesthesia | 16 | 20
  Lidocaine drip | 0 | 0

10. Secondary Outcome: Ventilator Free Days
Description: Number of inpatient hospital days patients did not require mechanical ventilation
Time Frame: Hospital discharge (up to 6 weeks post hospital admission)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 144 | 156
days | 30 [29 to 30] | 30 [29 to 30]

11. Secondary Outcome: ICU Free Days
Description: Number of inpatient hospital days patients did not require ICU level of care
Time Frame: Hospital discharge (up to 6 weeks post hospital admission)
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 144 | 156
days | 29 [26 to 30] | 28 [26 to 30]

12. Secondary Outcome: Hospital Free Days
Description: Number of days patients were not in the hospital during the first 30 days after admission
Time Frame: 30 days post admission
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 144 | 156
days | 20 [13 to 25] | 21 [13 to 25]

13. Secondary Outcome: Number of Patients Discharged From the Hospital With an Opioid Prescription
Description: Number of patients discharged from the hospital with an opioid prescription
Time Frame: Hospital discharge (up to 6 weeks post hospital admission)
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 144 | 156
Participants
  Any Opioid at discharge | 82 | 97
  Tramadol | 72 | 81
  Hydrocodone | 3 | 2
  Oxycodone | 10 | 15
  Codeine | 1 | 3
  Methadone | 0 | 0
  Fentanyl patch | 0 | 0
  Hydromorphone | 0 | 0
  Morphine | 1 | 0

14. Secondary Outcome: Number of Patients Who Reported Continued Pain Continued Post-traumatic Pain at 6 Months Post Admission
Description: Number of patients who reported continued pain at 6 months following trauma injury
Time Frame: 6 months post admission
Population: Data were not collected from 54 participants in the Usual Care arm and 44 in the Ketamine plus Usual Care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 100 | 102
Participants | 78 | 71

15. Secondary Outcome: Number of Patients Who Continue to Use Opioids at 6 Months Post Admission
Description: Number of patients who continue to use opioids
Time Frame: 6 months post admission
Population: Data were not collected from 54 participants in the Usual Care arm and 44 in the Ketamine plus Usual Care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 100 | 102
Participants | 11 | 11

16. Secondary Outcome: Post Traumatic Stress Disorder (PTSD) as Assessed by the PC-PTSD-5 Questionnaire
Description: The PC-PTSD-5 questionnaire asks the below 5 questions, and data are reported categorically as the number of participants who responded "yes" to each of the 5 questions. An answer of "yes" is indicative of a PTSD symptom, which is a worse outcome.
  1. In the past month, have you had nightmares about the events or thought about the events when you did not want to?
  2. In the past month, have you tried hard not to think about the events or went out of your way to avoid situations that reminded you of the events?
  3. In the past month, have you been constantly on guard, watchful, or easily startled?
  4. In the past month, have you felt numb or detached from people, activities, or your surroundings?
  5. In the past month, have you felt guilty or unable to stop blaming yourself or others for the events or any problems the events may have caused?
Time Frame: 6 months post admission
Population: These data were not collected from 78 participants in the Usual Care arm and 75 in the Ketamine plus Usual Care arm
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 69 | 78
Participants
  1. had nightmares about the events or thought about the events when you did not want to | 24 | 19
  2. tried hard not to think about the events or went out of your way to avoid situations | 41 | 44
  3. been constantly on guard, watchful, or easily startled | 42 | 47
  4. felt numb or detached from people, activities, or your surrounding | 37 | 36
  5. felt guilty or unable to stop blaming yourself or others | 24 | 23

17. Secondary Outcome: Risk of Future Opioid Abuse as Assessed by the Opioid Risk Tool (ORT)
Description: Total ORT score ranges from 0 to 26. A score of 3 or lower indicates low risk for future opioid abuse, a score of 4 to 7 indicates moderate risk for opioid abuse, and a score of 8 or higher indicates a high risk for opioid abuse.
Time Frame: Hospital discharge (about 1 to 6 weeks after admission)
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 124 | 129
Participants
  Low risk of future opioid abuse (score of 0-3) | 92 | 94
  Moderate risk of future opioid abuse (score of 4-7) | 13 | 25
  High risk of future opioid abuse (score of 8 or higher) | 19 | 10

18. Secondary Outcome: Health Status as Assessed by the Euro-QOL EQ-5D-3L Questionnaire (Mobility)
Description: For this item of the Euro-QOL EQ-5D-3L questionnaire, participants are asked to indicate their level of mobility by choosing a predefined category, and the data for this outcome are reported categorically as the number of participants who chose each category.
Time Frame: Hospital discharge (about 1 to 6 weeks after admission)
Population: These data were not collected from 27 participants in the Usual Care arm and 20 in the Ketamine plus Usual Care arm
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 124 | 129
Participants
  I have no problems walking | 39 | 31
  I have slight problems walking | 22 | 20
  I have moderate problems walking | 15 | 13
  I have severe problems walking | 13 | 17
  I am unable to walk | 35 | 48

19. Secondary Outcome: Health Status as Assessed by the Euro-QOL EQ-5D-3L Questionnaire (Self-Care)
Description: For this item of the Euro-QOL EQ-5D-3L questionnaire, participants are asked to indicate their level of self-care by choosing a predefined category, and the data for this outcome are reported categorically as the number of participants who chose each category.
Time Frame: Hospital discharge (about 1 to 6 weeks after admission)
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 124 | 129
Participants
  I have no problems washing or dressing myself | 42 | 37
  I have slight problems washing or dressing myself | 24 | 19
  I have moderate problems washing or dressing myself | 13 | 15
  I have severe problems washing or dressing myself | 5 | 7
  I am unable to wash or dress myself | 40 | 51

20. Secondary Outcome: Health Status as Assessed by the Euro-QOL EQ-5D-3L Questionnaire (Usual Activities)
Description: For this item of the Euro-QOL EQ-5D-3L questionnaire, participants are asked to indicate their ability to carry out usual activities by choosing a predefined category, and the data for this outcome are reported categorically as the number of participants who chose each category.
Time Frame: Hospital discharge (about 1 to 6 weeks after admission)
Population: These data were not collected from 27 participants in the Usual Care arm and 20 in the Ketamine plus Usual Care arm
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 124 | 129
Participants
  I have no problems doing my usual activities | 17 | 7
  I have slight problems doing my usual activities | 8 | 10
  I have moderate problems doing my usual activities | 5 | 9
  I have severe problems doing my usual activities | 2 | 4
  I am unable to do my usual activities | 92 | 99

21. Secondary Outcome: Health Status as Assessed by the Euro-QOL EQ-5D-3L Questionnaire (Pain/Discomfort)
Description: For this item of the Euro-QOL EQ-5D-3L questionnaire, participants are asked to indicate their level of pain/discomfort by choosing a predefined category, and the data for this outcome are reported categorically as the number of participants who chose each category.
Time Frame: Hospital discharge (about 1 to 6 weeks after admission)
Population: These data were not collected from 27 participants in the Usual Care arm and 20 in the Ketamine plus Usual Care arm
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 124 | 129
Participants
  I have no pain or discomfort | 25 | 16
  I have slight pain or discomfort | 34 | 32
  I have moderate pain or discomfort | 30 | 39
  I have severe pain or discomfort | 21 | 18
  I have extreme pain or discomfort | 14 | 24

22. Secondary Outcome: Health Status as Assessed by the Euro-QOL EQ-5D-3L Questionnaire (Anxiety/Depression)
Description: For this item of the Euro-QOL EQ-5D-3L questionnaire, participants are asked to indicate their level of anxiety/depression by choosing a predefined category, and the data for this outcome are reported categorically as the number of participants who chose each category.
Time Frame: Hospital discharge (about 1 to 6 weeks after admission)
Population: These data were not collected from 27 participants in the Usual Care arm and 20 in the Ketamine plus Usual Care arm
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 124 | 129
Participants
  I am not anxious or depressed | 70 | 74
  I am slightly anxious or depressed | 24 | 20
  I am moderately anxious or depressed | 11 | 15
  I am severely anxious or depressed | 6 | 7
  I am extremely anxious or depressed | 13 | 13

23. Secondary Outcome: Health Status as Assessed by the Euro-QOL EQ-5D-3L Questionnaire (Current Health)
Description: For this item of the Euro-QOL EQ-5D-3L questionnaire, participants are asked the question "How would you rate your health today?," and they respond with a score from 0 - 100, with a higher score indicating a better outcome.
Time Frame: Hospital discharge (about 1 to 6 weeks after admission)
Population: These data were not collected from 27 participants in the Usual Care arm and 20 in the Ketamine plus Usual Care arm
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 144 | 129
score on a scale | 70 [50 to 90] | 75 [50 to 80]

24. Secondary Outcome: Health Status as Assessed by the Euro-QOL EQ-5D-3L Questionnaire (Previous Experience)
Description: For this item of the Euro-QOL EQ-5D-3L questionnaire, participants are asked the question "Have you ever experience this kind of event?," and data are reported as the number of participants who responded "yes."
Time Frame: Hospital discharge (about 1 to 6 weeks after admission)
Population: These data were not collected from 27 participants in the Usual Care arm and 20 in the Ketamine plus Usual Care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 124 | 129
Participants | 82 | 77

25. Secondary Outcome: Health Status as Assessed by the Euro-QOL EQ-5D-3L Questionnaire (Mobility)
Description: as for outcome 18
Time Frame: 6 months post admission
Population: These data were not collected from 54 participants in the Usual Care arm and 44 in the Ketamine plus Usual Care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 100 | 102
Participants
  I have no problems walking | 50 | 47
  I have slight problems walking | 15 | 21
  I have moderate problems walking | 12 | 17
  I have severe problems walking | 9 | 8
  I am unable to walk | 14 | 9

26. Secondary Outcome: Health Status as Assessed by the Euro-QOL EQ-5D-3L Questionnaire (Self-Care)
Description: as for outcome 18
Time Frame: 6 months post admission
Population: These data were not collected from 54 participants in the Usual Care arm and 44 in the Ketamine plus Usual Care arm.
  1 participant in the Ketamine plus Usual Care arm did not complete the Self-Care section of the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 100 | 102
Participants
  I have no problems washing or dressing myself | 29 | 38
  I have slight problems washing or dressing myself | 12 | 10
  I have moderate problems washing or dressing myself | 16 | 14
  I have severe problems washing or dressing myself | 9 | 11
  I am unable to wash or dress myself | 34 | 28

27. Secondary Outcome: Health Status as Assessed by the Euro-QOL EQ-5D-3L Questionnaire (Usual Activities)
Description: as for outcome 20
Time Frame: 6 months post admission
Population: These data were not collected from 54 participants in the Usual Care arm and 44 in the Ketamine plus Usual Care arm.
  1 participant in the Usual Care arm did not complete the Usual Activities section of the Survey
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 100 | 102
Participants
  I have no problems doing my usual activities | 29 | 38
  I have slight problems doing my usual activities | 12 | 10
  I have moderate problems doing my usual activities | 16 | 14
  I have severe problems doing my usual activities | 9 | 11
  I am unable to do my usual activities | 34 | 28

28. Secondary Outcome: Health Status as Assessed by the Euro-QOL EQ-5D-3L Questionnaire (Pain/Discomfort)
Description: as for outcome 21
Time Frame: 6 months post admission
Population: These data were not collected from 54 participants in the Usual Care arm and 44 in the Ketamine plus Usual Care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 100 | 102
Participants
  I have no pain or discomfort | 31 | 25
  I have slight pain or discomfort | 17 | 21
  I have moderate pain or discomfort | 21 | 24
  I have severe pain or discomfort | 10 | 18
  I have extreme pain or discomfort | 21 | 14

29. Secondary Outcome: Health Status as Assessed by the Euro-QOL EQ-5D-3L Questionnaire (Anxiety/Depression)
Description: as for outcome 22
Time Frame: 6 months post admission
Population: These data were not collected from 54 participants in the Usual Care arm and 44 in the Ketamine plus Usual Care arm.
  2 participants in the Usual Care arm did not complete the Anxiety and Depression section in the survey.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 100 | 102
Participants
  I am not anxious or depressed | 50 | 53
  I am slightly anxious or depressed | 15 | 19
  I am moderately anxious or depressed | 11 | 13
  I am severely anxious or depressed | 4 | 2
  I am extremely anxious or depressed | 18 | 15

30. Secondary Outcome: Health Status as Assessed by the Euro-QOL EQ-5D-3L Questionnaire (Current Health)
Description: as for outcome 23
Time Frame: 6 months post admission
Population: These data were not collected from 54 participants in the Usual Care arm and 44 in the Ketamine plus Usual Care arm.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 100 | 102
score on a scale | 75 [60 to 90] | 80 [65 to 90]

31. Secondary Outcome: Health Status as Assessed by the Euro-QOL EQ-5D-3L Questionnaire (Previous Experience)
Description: as for outcome 24
Time Frame: 6 months post admission
Population: These data were not collected from 54 participants in the Usual Care arm and 44 in the Ketamine plus Usual Care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 100 | 102
Participants | 69 | 78

32. Secondary Outcome: Post Traumatic Stress Disorder (PTSD) as Assessed by the PC-PTSD-5 Questionnaire
Description: as for outcome 16
Time Frame: Hospital discharge (about 1 to 6 weeks after admission)
Population: These data were not collected from 74 participants in the Usual Care arm and 67 in the Ketamine plus Usual Care arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 77 | 82
Participants
  1. had nightmares about the events or thought about the events when you did not want to | 30 | 18
  2. tried hard not to think about the events or went out of your way to avoid situations | 35 | 49
  3. been constantly on guard, watchful, or easily startled | 36 | 43
  4. felt numb or detached from people, activities, or your surrounding | 24 | 31
  5. felt guilty or unable to stop blaming yourself or others | 19 | 25

33. Secondary Outcome: Pain as Assessed by Score on the Behavioral Pain Scale (BPS)
Description: BPS score ranges from 3-12, with higher scores indicating worse pain. This assessment is used in non-verbal participants.
Time Frame: Hospital discharge (up to 6 weeks post hospital admission)
Population: Data were not collected for this outcome measure
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 0 | 0

34. Secondary Outcome: Pain as Assessed by Average Score on the Defense and Veterans Pain Rating Scale (DVPRS)
Description: DVPRS scores were collected daily. For each participant, an average of the daily scores on the Defense and Veterans Pain Rating Scale was calculated. DVPRS scores range from 0 (no pain) to 10 (as bad as it could be, nothing else matters), with a higher score indicating a worse outcome.
Time Frame: From time of admission to time of discharge from hospital (about 1 to 6 weeks after admission)
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Ketamine Plus Usual Care | Usual Care
Number analyzed (Participants) | 144 | 156
score on a scale | 2.9 [1.6 to 4.3] | 2.5 [1.2 to 4.2]

ADVERSE EVENTS:
Time Frame: At time of Hospital discharge(up to 6 weeks post hospital admission)
Arm/Group | Ketamine Plus Usual Care | Usual Care
All-Cause Mortality (participants affected / at risk) | 1/144 | 6/156
Serious Adverse Events (participants affected / at risk) | 0/144 | 0/156
Other Adverse Events (participants affected / at risk) | 0/144 | 0/156

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-08-25): https://cdn.clinicaltrials.gov/large-docs/86/NCT04129086/Prot_SAP_000.pdf